CLINICAL TRIAL: NCT02679222
Title: Comparing the Ketogenic Effect of Coconut Oil and Different Medium-chain Triglycerides
Brief Title: Comparing the Ketogenic Effect of Coconut Oil and Different MCTs
Acronym: MCT-Coco
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2016-541
Record Dates: First submitted 2016-02-01; First posted 2016-02-10 (Estimated); Results first posted 2020-04-06 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-03

CONDITIONS: Healthy Adults
Keywords: Ketones; Coconut oil; Medium Chain Triglycerides
MeSH Terms: conditions — Ketosis | interventions — Coconut Oil; tricaprylin; tricaprin; Neprilysin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Supplementation (Experimental): Protocol involved seven separate but identical metabolic study days for each participant. the test substances were evaluated in random order: vehicle (Control) or 20 mL of the test oils (Coconut oil; tricaprin; tricaprylin; MCT [tricaprylin/tricaprin]; coconut oil + MCT [50:50]; Coconut oil + tricaprylin [50:50]) taken twice, once at breakfast and once at mid-day.
  Interventions: Dietary Supplement: Coconut oil; Dietary Supplement: Coconut oil + MCT; Dietary Supplement: MCT; Dietary Supplement: Coconut oil + tricaprylin; Dietary Supplement: Tricaprylin; Dietary Supplement: Tricaprin; Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Coconut oil — 20 g of coconut oil
  Other Names: Coco
Dietary Supplement: Coconut oil + MCT — 10 g of coconut oil + 10 g of MCT (60 of C8 + 40 of C10)
  Other Names: Coco+MCT
Dietary Supplement: MCT — 20 g of MCT (60 of C8+40 of C10)
Dietary Supplement: Coconut oil + tricaprylin — 10 g coconut oil + 10 g tricaprylin
  Other Names: Coco+C8
Dietary Supplement: Tricaprylin — 20 g tricaprylin
  Other Names: C8
Dietary Supplement: Tricaprin — 20 g tricaprin
  Other Names: C10
Dietary Supplement: Control — No supplement taken on this visit
  Other Names: CTL

SUMMARY:
The aim of this study is to compare the ketogenic effect of coconut oil and three MCT oils (60-40 , tricaprylin and triheptanoate) on the production of ketones in healthy adults. Each oil are evaluated individually or in combination over a 8h-period during which repeated blood sampling is performed.

DETAILED DESCRIPTION:
The study is composed of eight successive visits. Each visit consists of the consumption of one individual oil or a mixture of oils (20 g of coconut oil or 10 g of coconut oil + 10 g of MCT 60-40 or 20 g MCT 60-40 or 10 g coconut oil + 10 g tricaprylin or 20 g tricaprylin or 10 g coconut oil + 10 g triheptanoate or 20 g triheptanoate) and a 8h follow-up during which repeated blood samples are taken for laboratory analysis (plasma beta-hydroxybutyrate, acetoacetate, glucose, free fatty acids, triglycerides, total cholesterol, lactate and insulin).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult over 18 y old.

Exclusion Criteria:

* Fasting plasma glucose ≥7.0 mM (diabetics or pre-diabetics);
* Smoking
* Clinically-significant gastro-intestinal disease/conditions.
* Clinically-significant liver disease/dysfunction.
* Clinically-significant cardiac disease/conditions.
* Clinically-significant abnormal coagulation.
* Taking a medication that could affect lipid and glucose metabolism
* Hypertension
* Pregnancy or breastfeeding
* Exercising more than 3 times a week

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Cunnane, PhD, Principal Investigator — CSSS-IUGS - CIUSSS de L'Estrie - CHUS - Université de Sherbrooke
Locations (1):
- Research Centre on Aging (CSSS-IUGS - CIUSSS de l'Estrie - CHUS), Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Supplementation
Started | 10
Completed | 9
Not Completed | 1
Not completed — No time for project | 1

BASELINE CHARACTERISTICS:
Arm/Group | Supplementation
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 9
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 24 (3)
Glucose [Mean (Standard Deviation); unit: mmol/L] | 4.3 (0.2)
Ketones [Mean (Standard Deviation); unit: µmol/L] | 90 (61)

OUTCOME MEASURES:

1. Primary Outcome: Plasma Ketone Concentrations
Description: Total ketones = Plasma acetoacetate (µmol/L) + beta-hydroxybutyrate (µmol/L) measured over a 8 hour period (i.e. daily mean).
  Samples are taken every 30 minutes on a 8 hours period. The mean is reported here.
Time Frame: 8 hours
Measure: Mean (Standard Deviation); unit: µmol/L
Groups:
- Control: vehicle (Control) taken twice, once at breakfast and once at mid-day.
  Control: No supplement taken on this visit
- Medium Chain Triglyceride: 20 mL of MCT taken twice, once at breakfast and once at mid-day.
  MCT: 20 g of MCT (60 of C8+40 of C10)
- Tricaprin: 20 mL of MCT tricaprin taken twice, once at breakfast and once at mid-day.
  Tricaprin: 20 g tricaprin
- Tricaprylin: 20 mL of tricaprylin taken twice, once at breakfast and once at mid-day.
  Tricaprylin: 20 g tricaprylin
- Coconut Oil: 20 mL of Coconut oil taken twice, once at breakfast and once at mid-day.
  Coconut oil: 20 g of coconut oil
- Coconut Oil + MCT: 20 mL of coconut oil + MCT taken twice, once at breakfast and once at mid-day.
  Coconut oil + MCT: 10 g of coconut oil + 10 g of MCT (60 of C8 + 40 of C10)
- Coconut Oil + Tricaprylin: 20 mL of Coconut oil + tricaprylin [50:50]) taken twice, once at breakfast and once at mid-day.
  Coconut oil + tricaprylin: 10 g coconut oil + 10 g tricaprylin
Arm/Group | Control | Medium Chain Triglyceride | Tricaprin | Tricaprylin | Coconut Oil | Coconut Oil + MCT | Coconut Oil + Tricaprylin
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 9
µmol/L | 69 (92) | 294 (85) | 109 (41) | 363 (109) | 107 (97) | 141 (39) | 235 (79)

2. Secondary Outcome: Plasma Acetoacetate/Beta-hydroxybutyrate Ratio
Description: Plasma ratio of acetoacetate (µmol/L)/ beta-hydroxybutyrate (µmol/L) measured over a 8 hour period (i.e area-under-the-curve over 8 hours).
Time Frame: 8 hours
Measure: Mean (Standard Deviation); unit: Ratio
Groups:
- Tricaprin: 20 mL of MCT tricaprintaken twice, once at breakfast and once at mid-day.
  Tricaprin: 20 g tricaprin
- Coconut Oil +t Tricaprylin: 20 mL of Coconut oil + tricaprylin [50:50]) taken twice, once at breakfast and once at mid-day.
  Coconut oil + tricaprylin: 10 g coconut oil + 10 g tricaprylin
Arm/Group | Control | Medium Chain Triglyceride | Tricaprin | Tricaprylin | Coconut Oil | Coconut Oil + MCT | Coconut Oil +t Tricaprylin
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 9
Ratio | 7.7 (3.2) | 6.9 (1.5) | 7.7 (1.1) | 5.9 (1.0) | 9.5 (2.9) | 8.4 (1.3) | 8.1 (2.2)

ADVERSE EVENTS:
Time Frame: 7 visits of 8 hours
Arm/Group | Supplementation
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes